CLINICAL TRIAL: NCT03006224
Title: The Effects of Secondary Smoking to Intraoperative Arterial Oxygen Tension During One Lung Ventilation in Lobectomy
Brief Title: The Effects of Secondary Smoking During One Lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ahmet Selim Ozkan, M.D., Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Asozkan-5
Record Dates: First submitted 2016-12-22; First posted 2016-12-30 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Smoking; Oxygen Deficiencies
Keywords: secondary smoking; one lung ventilation; arterial oxygen tension; lobectomy
MeSH Terms: conditions — Smoking; Hypoxia | interventions — One-Lung Ventilation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group S (non smoking and secondary smoking) (Active Comparator): I want to see the effects of seconder smoking to intraoperative arterial oxygen tension during one lung ventilation for lobectomy surgery.
  Interventions: Other: One Lung Ventilation
- Group SS (secondary smoking) (Active Comparator): I want to see the effects of seconder smoking to intraoperative arterial oxygen tension during one lung ventilation for lobectomy surgery.
  Interventions: Other: One Lung Ventilation

INTERVENTIONS:
Other: One Lung Ventilation

SUMMARY:
Smoking and perhaps secondary smoking is associated with many perioperative and postoperative complications, especially respiratory events. Hypoxemia and airway damage can be associated with secondary smoking. The aim of study is to predict the incidence of hypoxemia and airway damage during one lung ventilation for lobectomy.

DETAILED DESCRIPTION:
Sixty patients undergoing lobectomy using one lung ventilation by double lumen tube will be included in this study. These patients will be divided into 2 groups. Groups S which will be included non smoking and secondary smoking and group SS which will be included secondary smoking ( smoking near him more than 10 cigarettes per day fore more than 5 years). Intra and postoperative arterial oxygen tension, arterial carbon dioxide tension and intraoperative peak airway pressure will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Sixty patients undergoing lobectomy using one lung ventilation by double lumen tube, ASA physical status 2 and 3.

Exclusion Criteria:

* Recent chest infection, morbid obesity, renal, hepatic and ischemic hearts disease, asthma.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
arterial oxygen tension | From beginning of Anesthesia to 1st day of surgery
arterial carbon dioxide tension | From beginning of Anesthesia to 1st day of surgery
intraoperative peak airway pressure | during intraoperative ventilation

IPD SHARING:
Plan to Share IPD: Undecided